CLINICAL TRIAL: NCT01569737
Title: Prospective Multicenter Observational Study to Assess Clinical Follow-up and Outcomes of Pregnancies Exposed to Ella
Brief Title: Clinical Follow-up and Outcomes of Pregnancies Exposed to Ella
Acronym: ellipseII
Status: Completed | Type: Observational
Sponsor: HRA Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2914-012
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Emergency Contraception
Keywords: ella; ulipristal acetate; pregnancy; emergency contraception
MeSH Terms: interventions — ulipristal acetate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ella
  Interventions: Drug: ella

INTERVENTIONS:
Drug: ella — ella, single intake, tablet 30mg

SUMMARY:
The study is aimed at assessing the clinical follow-up and the outcomes of pregnancies exposed to ella, whether due to failure of the emergency contraception or inadvertent exposure during pregnancy.

ELIGIBILITY:
* Pregnant women, exposed to ella during the menstrual cycle in which the pregnancy started (treatment failure) or at any time during pregnancy (inadvertent exposure during pregnancy)
* Adolescents and/or adults in the USA, depending on the respective State law

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women who have been exposed to ella during the menstrual cycle in which the pregnancy started or at any time during pregnancy will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Fine, MD, Principal Investigator — Planned Parenthood Gulf Coast
Locations (1):
- Planned Parenthood Federation of America, Inc, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ella-exposed pregnant women were recruited either by Health Care Professionals at Family Planning Clinics or through web-based self enrollment between November 2014 and December 2017.
  The first participant was enrolled on November 18, 2014 and the last participant was enrolled December 12, 2017.
Period: Overall Study
Arm/Group | Ella
Started | 98
Completed | 95
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ella
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Outcome was not known for 3 patients, thus not included in the Analysis population.
  years
    number analyzed (Participants) | 95
    (all) | 26.6 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 98
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Analysis includes all patients for whom values were known.
  kg/m^2
    number analyzed (Participants) | 95
    (all) | 26.7 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Assessed Pregnancy Outcomes
Description: Live birth outcomes:
  Healthy baby; Congenital anomaly: a baby born with a congenital anomaly; Neonatal death: a newborn who died during the first 28 days of life; Preterm birth: a baby born at less than 37 weeks of gestational age;
  Pregnancy loss outcomes:
  Ectopic pregnancy: implantation of the fertilized egg and pregnancy development in a location outside the uterus and attempt to develop in this location; Spontaneous abortion: early fetal death (i.e. less than 20 completed weeks of gestation);
  Fetal death:
  Intermediate fetal death (between greater than 20 and less than 28 completed weeks of gestation); Late fetal death (greater or equal to 28 completed weeks of gestation);
  Induced abortions can be either:
  An induced abortion for non-medical reason; An induced abortion for medical reasons (termination of pregnancy for fetal anomaly, or for other pregnancy or maternal health complications)
Time Frame: up to 9 months after pregnancy diagnosis
Population: Pregnancy outcomes were described for pregnancies with known outcome (patients with missing outcomes and patients lost to follow-up were excluded from the descriptive analyses).
Measure: Count of Participants; unit: Participants
Arm/Group | Ella
Number analyzed (Participants) | 95
Participants
  Healthy Live Births | 1
  total prevalence congenital anomalies | 0
  Ectopic Pregnancies | 1
  Spontaneous abortion | 0
  Fetal Deaths | 0
  Induced Abortions for non-medical reasons | 93
  Induced Abortions for medical reasons | 0
  Maternal Deaths | 0

ADVERSE EVENTS:
Time Frame: Adverse events were not collected in the context of this Phase IV observational study.
Description: When applicable, Individual Case Safety Reports were reported to Health Authorities on an expedited basis according to current regulation (no later than 15 calendar days from receipt).
  Unintended pregnancy reports (i.e. reports of pregnancies inadvertently exposed to ella without outcome data or with normal outcome) are considered as not serious by the company.
  Reports of the aggregate data concerning pregnancies were compiled and submitted to Health Authorities via PSUR.
Arm/Group | Ella
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This was an observational study only, thus we were limited to the outcomes reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Study protocol signed by the PI, (i) sponsor owns the study data (ii) HCP agrees that the results of the study may be used for the purposes of publications, and information for medical and pharmaceutical professionals (iii) if sponsor publishes the study results within 24-month, PI may elect to serve as co-authors, and following publication, will be permitted to present the results of such publications in symposia.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT01569737/SAP_000.pdf
  • Study Protocol and Informed Consent Form (2015-03-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT01569737/Prot_ICF_001.pdf